CLINICAL TRIAL: NCT01812577
Title: Evaluation of the Analgesic Efficacy of the Ultrasound Guided Thoracic Paravertebral Block for Percutaneous Radiofrequency Ablation of Liver Lesions
Brief Title: Paravertebral Block for Percutaneous Radiofrequency Ablation of Liver Lesions
Acronym: TPVB
Status: Completed | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Massimiliano Carassiti, MD, Campus Bio-Medico University
Other Study IDs: CarGal
Record Dates: First submitted 2013-03-08; First posted 2013-03-18 (Estimated); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Liver Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Thoracic paravertebral block (TPVB): Twenty patients receiving thoracic paravertebral block at level of T7, before the interventistic procedure.
- Deep Sedation (DS): Twenty patients receiving local and intravenous anesthesia during the procedure.

SUMMARY:
Percutaneous radiofrequency ablation of liver lesions causes patients acute pain during and after the procedure. During the procedure patients need deep sedation and cannot be collaborative. Furthermore post-operative analgesia is necessary. The aim of this study is to evaluate if the ultrasound-guided paravertebral block (TPVB)with a single injection can provide anesthesia and post-operative analgesia in these patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate if single injection TPVB, ultrasound guided, ENS assisted, is advantageous compared to deep sedation (DS)in patients undergoing percutaneous radiofrequency ablation of liver lesions with respect to post-operative analgesia (at rest and in movement)and vomiting. Furthermore we collect data on operator and patient satisfaction.

In this study patients are randomly divided into two groups (20 patient each): TPVB and DS. In TPVB group the block is performed in lateral position at level of T7 with bupivacaine 5mg/ml. In DS group the procedure is conducted under local and intravenous anesthesia, and a post-operative analgesia is assigned. Data on patient, on procedures (duration, number and position of lesions etc.), complications with the anesthesiological technique are collected. The intensity of post-operative pain is assessed at 3-6-12 and 24 hours after procedure in both group using VRS pain scale at rest and in movement. Any concomitant event like nausea, vomiting, respiratory complications etc are recorded.

ELIGIBILITY:
Inclusion Criteria:

* written consent ASA I-III

Exclusion Criteria:

* allergy to local anesthetic infection in the site of planned injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study 40 patients undergoing elective procedure of radiofrequency ablation of liver lesions are enrolled after written informed consent is obtained.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Intensity of postoperative pain after radiofrequency ablation of liver lesion | first 24 post-operative hours
  Intensity of postoperative pain after radiofrequency ablation of liver lesion is evaluated in both groups using VRS of pain at rest and in movement after 3-6-12-24 hours from procedure.

SECONDARY OUTCOMES:
Incidence of complications | From procedure to 24 hours
  We record immediate complication such as PNX, vascular puncture etc, and post-operative complications such as nausea, vomiting, hypotension, etc, in both groups
Consumption of post-operative opioid | Within 24 post-operative hours
  We evaluate if there is differences in consumption of opioid in the two groups

OTHER OUTCOMES:
Satisfaction of patient and of the operator | From the procedure to 24 hours later.
  We collect data on operator satisfaction during the procedure, and patients satisfaction at 24 hours after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Carassiti, MD, Principal Investigator — Campus Bio Medico
Locations (1):
- Campus Bio-Medico, Rome, Italy/RM, Italy

REFERENCES:
- [Background] Hara K, Sakura S, Nomura T, Saito Y. Ultrasound guided thoracic paravertebral block in breast surgery. Anaesthesia. 2009 Feb;64(2):223-5. doi: 10.1111/j.1365-2044.2008.05843.x. No abstract available. PMID 19143711
- [Background] Renes SH, Bruhn J, Gielen MJ, Scheffer GJ, van Geffen GJ. In-plane ultrasound-guided thoracic paravertebral block: a preliminary report of 36 cases with radiologic confirmation of catheter position. Reg Anesth Pain Med. 2010 Mar-Apr;35(2):212-6. doi: 10.1097/aap.0b013e3181c75a8b. PMID 20301827